CLINICAL TRIAL: NCT05818839
Title: Biomechanical Properties and Their Association With Balance and Functional Mobility in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Ilke KARA (Other)
Responsible Party: Sponsor-Investigator, Ilke KARA, Co-Investigator, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Other Study IDs: BEU-CP-01
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Cerebral Palsy
Keywords: postural balance; muscle properties; mobility; paralysis; children
MeSH Terms: conditions — Cerebral Palsy; Paralysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UCP: Children diagnosed with unilateral spastic cerebral palsy
- TyD: Typically developing children

SUMMARY:
This study aimed to investigate the differences in the biomechanical properties of the dorsal trunk and lower extremity muscles of children with unilateral spastic cerebral palsy compared with their typically developing peers, and the effect of these biomechanical properties on balance and functional mobility performance.

ELIGIBILITY:
Inclusion criteria for unilateral spastic cerebral palsy were:

* aged between 4 and 12 years,
* spasticity level MAS≤2,
* mental level sufficient to understand commands given,
* and ambulation without the use of an orthosis or other device. In addition, children had to be GMFCS level I or II.

Exclusion criteria were:

* a history of spinal surgery or spinal orthosis use,
* uncorrected vision or hearing problems,
* severe epileptic seizures,
* lower extremity contractures,
* botulinum toxin A injection in the previous six months,
* lower extremity surgery in less than one year,
* use of pharmacological agents that affect muscle tone,
* and poor cooperation.

Inclusion criteria for controls were:

* aged between 4 and 12 years,
* no neurological or orthopaedic diagnosis,
* no known systemic problems,
* normal vision and hearing,
* and a mental level sufficient to understand the commands given.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children diagnosed with unilateral spastic cerebral palsy (GMFCS level I-II, spasticity level MAS ≤ 2) and their age-matched typically developing peers.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
The Pediatric Balance Scale | Baseline
  The Pediatric Balance Scale assesses functional balance in three categories: self-care, mobility and social function, using 14 items. Each item is scored from 0 (indicating low function) to 4 (indicating highest function), with a maximum score of 56 points. A higher score indicates better balance.
Trunk Control Measurement Scale | Baseline
  The TCSM was used to assess seated trunk balance and consisted of 15 items. Each item was scored from 0 to 3, with 0 indicating inability to perform the task and 3 indicating the full performance of the item. A high score indicated good trunk control
2-Minute Walk Test | Baseline
  The children were asked to walk at a normal pace, without running, and the distance they walked for 2 minutes was recorded.
Timed Up and Go Test | Baseline
  The children were seated with their feet in full contact with the floor, in a chair with back support only, and with their hip and knee joints at 90 degrees. On the start command, they were asked to walk 3 metres to the wall at a pace they felt comfortable with and then sit back down in the chair.
Muscle tone (Hz) | Baseline
  The muscle tone which is a biomechanical property of the muscles evaluated with a portable hand-held myotonometer. This myotonometer (MyotonPRO - Tallinn, Estonia) is non-invasive and provides a quantitative assessment of a muscle's biomechanical properties. The MyotonPRO applies a short-intensity mechanical impulse on the skin overlying the muscle or facia. The tissue's response then generates a signal that is recorded, and an internal software program produces an acceleration graph.
Stiffness (N/m) | Baseline
  The stiffness which is a biomechanical property of muscles will be evaluated with a portable hand-held myotonometer. This myotonometer (MyotonPRO - Tallinn, Estonia) is non-invasive and provides a quantitative assessment of a muscle's biomechanical properties. The MyotonPRO applies a short-intensity mechanical impulse on the skin overlying the muscle or facia. The tissue's response then generates a signal that is recorded, and an internal software program produces an acceleration graph.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Okan University, Istanbul, Turkey (Türkiye)